CLINICAL TRIAL: NCT00683813
Title: Randomized Trial of a Cardiac Rehabilitation Program Delivered Remotely Through the Internet
Brief Title: Trial of a Cardiac Rehabilitation Program Delivered Remotely Through the Internet
Acronym: vCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Scott Lear, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38390
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Cardiovascular Disease
Keywords: cardiac rehabilitation; telehealth; Internet
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UC (No Intervention): usual care
- vCRP (Experimental)
  Interventions: Behavioral: vCRP

INTERVENTIONS:
Behavioral: vCRP — The vCRP includes online intake forms, one-on-one chat sessions with vCRP nurse, dietitian and exercise specialist, data collection (exercise heart rate, blood pressure, glucose- if diabetic), peer-support group chat sessions, ask-an-expert chat sessions, education, progress reports and online resources. VCRP patients will receive access to the website, a heart rate monitor and a blood pressure monitor and trained in their use. The heart rate monitors allow for exercise heart rate data to be stored and downloaded to their home computer and then uploaded to the vCRP webserver. The exercise data will be reviewed weekly. A letter to the patient's primary care physician will be sent to outline the vCRP intervention, the treatment algorithms to be used and indicate under what circumstances the vCRP nurse and/or patient may contact them with regards to their management. After the 4 month intervention, patients will be discharged into the care of their primary care physician.
  Arms: vCRP

SUMMARY:
Cardiac rehabilitation programs (CRP) are a proven treatment for those with ischemic heart disease (IHD). These programs have been demonstrated to improve adherence to regular physical activity, a healthy diet and smoking cessation, as well as modify risk factors for IHD such as hypercholesterolemia, hypertension, obesity and type 2 diabetes. In addition, CRP are cost effective and can result in a 25% reduction in reoccurrence of mortality. Despite the known benefits of CRP, as little as 10% to 25% of eligible patients attend these programs. One of the main barriers to attendance is proximity to a CRP, as the majority of these programs are limited to hospitals in large urban areas. However, cardiovascular diseases do not discriminate by geography, resulting in a geographic inequity of care for patients living in rural, remote and smaller urban/sub-urban centres. Currently there are no CRP specifically designed for patients in rural and remote areas. The use of the Internet may present itself as a viable alternative. We have recently completed a pilot study of a virtual CRP (vCRP) that demonstrated significant improvements in exercise capacity and risk factors. This investigation will study the vCRP in a group of IHD patients who do not have access to hospital-based CRP.

Hypotheses A. Participation in a 4 month Internet-based cardiac rehabilitation program will result in significant improvements in exercise capacity compared to usual care, in patients with diagnosed IHD.

B. Participation in a 4 month Internet-based cardiac rehabilitation program will result in significant improvements in exercise capacity after one year compared to usual care, in patients with diagnosed IHD.

Study Population Men and women over 18 years will be identified from consecutive in-patients of the British Columbia Provincial Heart Centre at St. Paul's Hospital in Vancouver who reside in either the Northern Interior or Coast Garibaldi health areas. Patients will be eligible if they have IHD, Internet access, no previous experience with cardiac rehabilitation and no physical limitations to exercise. A total of 74 patients (37 per group) will be recruited and randomized to either usual care, or a 4 month 'virtual' cardiac rehabilitation program delivered via the Internet.

Usual Care Group Patients randomized to usual care will be provided with simple guidelines for safe exercising and healthy eating habits, and return to the care of their primary care physician. Patients will return at 4 and 16 months later for outcome assessment. There will be no contact between the study personnel and usual care patients for the duration of the study, nor will there be any attempt to control the level of patient care.

Intervention The vCRP has been developed to mimic hospital-based CRP and includes online intake forms, one-on-one chat sessions with vCRP nurse, dietitian and exercise specialist, data collection (exercise heart rate, blood pressure, glucose- if diabetic), peer-support group chat sessions, ask-an-expert chat sessions, education, progress reports and online resources. Upon randomization to the intervention, patients will receive access to the website, a heart rate monitor and a blood pressure monitor and trained in their use. The heart rate monitors allow for exercise heart rate data to be stored and downloaded to their home computer and then uploaded to the vCRP webserver. The exercise data will be reviewed weekly. A letter to the patient's primary care physician will be sent to outline the vCRP intervention, the treatment algorithms to be used and indicate under what circumstances the vCRP nurse and/or patient may contact them with regards to their management. Patients will receive one-on-one counselling by the nurse, dietitian and exercise specialist via chat sessions at 3 to 4 week intervals. After the 4 month intervention, patients will be discharged into the care of their primary care physician.

Outcomes Participants will be assessed at baseline, 4 and 16 months for risk factors and lifestyle behaviours. The primary outcomes will be the change in exercise capacity as between the two groups from baseline to 4 months, and from baseline to 16 months. Exercise capacity will be assessed as total time on a symptom-limited exercise stress test.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women admitted for an IHD event (acute coronary syndrome or revascularization procedure) who are at low or moderate risk.91
2. Regular Internet access (home, work or other environment).
3. Over 18 years of age.
4. Permission of the attending physician.
5. Able to read, write and understand English without difficulty.
6. No physical limitations to regular activity.

Exclusion Criteria:

1. Previous experience with a cardiac rehabilitation program.
2. Patients with depression, uncontrolled diabetes and other significant co-morbidities that may interfere with effective IHD management.
3. Those patients, who in the mind of the attending physician, are unsuitable for participation.
4. Those unable to provide informed consent.
5. Pregnant women.
6. High-risk patients for safety considerations (future studies will include high-risk patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
exercise capacity as reported in total time on the exercise test using the BRUCE protocol | 16 months

SECONDARY OUTCOMES:
anthropometry | 4 months
blood lipids | 4 months
fasting blood glucose | 4 months
physical activity | 4 months
diet | 4 months
smoking status | 4 months
healthcare utilization | 16 months
exercise capacity | 4 months
anthropometry | 16 months
fasting blood glucose | 16 months
diet | 16 months
blood lipids | 16 months
physical activity | 16 months
smoking | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Lear, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Lear SA, Singer J, Banner-Lukaris D, Horvat D, Park JE, Bates J, Ignaszewski A. Randomized trial of a virtual cardiac rehabilitation program delivered at a distance via the Internet. Circ Cardiovasc Qual Outcomes. 2014 Nov;7(6):952-9. doi: 10.1161/CIRCOUTCOMES.114.001230. Epub 2014 Sep 30. No abstract available. PMID 25271050
- [Derived] Lear SA, Singer J, Banner-Lukaris D, Horvat D, Park JE, Bates J, Ignaszewski A. Improving access to cardiac rehabilitation using the internet: a randomized trial. Stud Health Technol Inform. 2015;209:58-66. PMID 25980706